CLINICAL TRIAL: NCT06381999
Title: Initial Assessment of the Validity and Inter-Rater Reliability for Early Recognition of Spasticity Using the Decision Tree Tool
Brief Title: Validity and Inter-rater Reliability for Early Recognition of Spasticity Using the Decision Tree Tool
Acronym: I-REFER
Status: Completed | Type: Observational
Sponsor: Merz Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Organization: Merz Pharmaceuticals GmbH (Industry)
Other Study IDs: M602011083
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Post-stroke Spasticity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the validity and Inter-rater reliability for early recognition of spasticity by nurses and physiotherapists using the decision tree tool.

DETAILED DESCRIPTION:
The Spastic Movement Disorder (SMD) Decision Tree was designed as a tool to aid nurses, therapists and other healthcare professions recognize potential signs of disabling spasticity in the upper limb of post-stroke patients. The present study assesses validity and inter-rater reliability of the SMD Decision Tree comparing nurses and therapists with gold-standard procedure performed by rehabilitation doctors. Agreement was tested for "referral to specialist indicated" and "no referral to specialist indicated".

ELIGIBILITY:
Inclusion Criteria:

* Participants with a first sub-acute and chronic infarction of the middle cerebral artery / basal ganglia hemorrhage longer than four weeks after the event
* Between 18-80 years old
* Preserved insight and judgment capacity
* Adequate language and task comprehension, attention span for 15 minutes

Exclusion Criteria:

* Participants with other neurological disorders
* Participants who received BoNT-A treatment < 3 months before inclusion
* Reduced vigilance and attention span (less than 15 minutes)
* Participants with adult representation
* Participants with severe language impairment / impairment of movement and action sequences

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male, Female, and Diverse were eligible.
Study Population: Study participants are post-stroke survivors and patients of the Gailtal Clinic in Hermagor.
  Participants were either sub-acute in-patients as part of the post-stroke rehabilitation program or chronic out-patients.
  Participants are recruited using consecutive participant sampling. All sub-acute patients in the rehabilitation ward who fulfill inclusion criteria and agree to participate are enrolled. Additionally, chronic patients scheduled for botulinum toxin injections on the study day are also enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Assessment of the level of agreement between the nurse group and gold-standard group (trained, specialized physicians) in their decision for toxin treatment referral | Day 1-2
  Nurses use the 3 domains of the SMD Decision Tree (passive/active movement, pain) to determine potential disabling spasticity indicated for referral to a rehabilitation specialist. Specialized physicians use standard clinical procedure to detect disabling spasticity.

SECONDARY OUTCOMES:
Assessment of the level of agreement between the physiotherapist and/or occupational therapist group and gold-standard group (trained, specialized physicians) in their decision for toxin treatment referral | Day 1-2

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Therapeutics
Locations (1):
- Gailtal-Klinik, Hermagor, Austria

IPD SHARING:
Plan to Share IPD: No